CLINICAL TRIAL: NCT02403518
Title: A Prospective, Multi-National, Post-Marketing Study of the Clinical Outcomes of Wireless Neuromodulation Via the Freedom Spinal Cord Stimulation (SCS) System for the Management of Chronic Back and Leg Pain
Brief Title: Clinical Outcomes of the Freedom Spinal Cord Stimulation (SCS) System for the Management of Chronic Back and Leg Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Curonix LLC (Industry)
Collaborators: Amphia ziekenhuis, Oosterhout, The Netherlands (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0071
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Low Back Pain; Pain in Leg, Unspecified

ARMS (3):
- Back Pain Only (Active Comparator): Pain localized to the low back or buttocks.
  Interventions: Device: Freedom Spinal Cord Stimulator System
- Leg Pain Only (Active Comparator): Pain localized to unilateral pain of the leg (thigh, knee, calf, or foot).
  Interventions: Device: Freedom Spinal Cord Stimulator System
- Back and Leg Pain (Active Comparator): Pain localized to both the low back and legs (back, buttocks, thigh, knee, calf, or foot).
  Interventions: Device: Freedom Spinal Cord Stimulator System

INTERVENTIONS:
Device: Freedom Spinal Cord Stimulator System
  Other Names: Freedom-4 SCS System; Freedom-4A SCS System; Freedom-8A SCS System

SUMMARY:
This study evaluates the Freedom SCS (spinal cord stimulation) System for the treatment of chronic back and leg pain. Patients who have been diagnosed with failed back surgery syndrome (FBSS) will receive a stimulator device for treatment of their pain.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate Freedom SCS candidate as affirmed by study investigator
* Candidate has a stable spine not suitable for further surgery as confirmed by physician
* 18 years of age or older (no upper age limit)
* Diagnosis of failed back surgery syndrome (FBSS) characterized by chronic, intractable pain of the legs, back, or both legs and back
* At least 6 months since last surgical procedure on the spine
* Average score of 60mm or greater on a VAS scale (Scale of 0 to 100, where 0 equals no pain and 100 equals worst possible pain)
* Pain duration of at least 6 months
* Expected lifespan of at least two years
* Able to comply with study requirements
* Gives informed consent for study participation

Exclusion Criteria:

* A consistent VAS score of 100 over the past 24 hours as established at Visit 1
* A co-existing condition that could increase the risk of SCS implantation (e.g., severe cardiac or respiratory disorders, coagulation disorder) or planned surgery within the study duration that could be compromised by SCS (e.g., diathermy)
* Pregnant or planning to become pregnant
* Known or suspected substance abuse within the last 2 years
* Major psychiatric disorder (untreated or refractory to treatment) in the investigators opinion
* Cognitive and/or behavioral issues that could impair study participation, (e.g., unreliability; defective memory; noncompliance in taking medications or keeping appointments; or impaired orientation to time, place, and events)
* Documented allergy to Freedom SCS material components
* Co-existing pain condition or participation in another clinical study that could confound the results of this study
* History of another implanted medical device (e.g., explanted spinal cord stimulator, peripheral nerve stimulation, sacral nerve stimulator, pacemaker, or intrathecal drug delivery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Percentage of pain relief experienced in the area of pain identified at baseline compared to 12 months post full implant of the Freedom SCS system. | 12 months
  Self reported pain intensity measured by the Visual Analog Scale (VAS)
Incidence and severity of device related adverse events during the study. | Up to 12 months

SECONDARY OUTCOMES:
To assess compliance data to indicate usability of the device. | 12 Months
  Questionnaire
To assess the implanters' experience with the device. | Average of 7 days after implant
  Questionnaire
Patient satisfaction with treatment. | 12 Months
  Questionnaire
Reduced visits to health care institutes for chronic back and leg pain. | 12 Months
  Questionnaire
Improved work status. | 12 Months
  Questionnaire
Improved quality of life function via the ODI and EQ-5D questionnaires | 12 Months
  ODI and EQ-5D Questionnaires
Reduction in use of analgesics | 12 Months
Reduced operating theater time | Average of 7 days after implant
  Review of hospital records
Reduced skin to skin time | Average of 7 days after implant
  Review of hospital records
Reduced skin to fluoroscope time | Average of 7 days after implant
  Review of hospital records
To monitor non-device and non-SCS-related adverse events | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Greg Jansen, Principal Investigator — Amphia ziekenhuis Oosterhout
Locations (1):
- Amphia Ziekenhuis, Oosterhout, North Brabant, Netherlands